CLINICAL TRIAL: NCT00103376
Title: VELCADE® (Bortezomib) for Injection Therapy for Early Relapsed Prostate Cancer
Brief Title: Bortezomib With or Without Hormone Therapy in Treating Patients With Relapsed Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000406013; MUSC-031218; MUSC-HR-11357
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Bortezomib; Gonadotropin-Releasing Hormone; Androgen Receptor Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A: Velcade (Experimental): Patient will complete Part A (Velcade only). If the patient has a complete response, he will come off study. If the patient has progressive disease, he will start Part B (Velcade + antiandrogen). If the patient has a partial response or stable disease, he will start Part B after at least a 7-day break.
  Interventions: Drug: Velcade
- Part B: Velcade+LH-RH antagonist+Androgen receptor antagonist (Experimental): Patient will start Part B after completing Part A or may be enrolled to part B only.
  Interventions: Drug: Velcade; Drug: LH-RH Agonist; Drug: Androgen Receptor Antagonists

INTERVENTIONS:
Drug: Velcade — Part A: 1.3 mg/m2 administered on days 1, 4, 8 and 11 followed by 10 days rest. A second cycle will be given at the same schedule. Cycle 3 will include 3 weekly injections.
  Part B: 1.3mg/m2 administered weekly for 3 weeks followed by 1 week break
  Other Names: bortezomib
Drug: LH-RH Agonist — given as a 3 month depo-injection
  Arms: Part B: Velcade+LH-RH antagonist+Androgen receptor antagonist
Drug: Androgen Receptor Antagonists — given orally daily for 3 months
  Arms: Part B: Velcade+LH-RH antagonist+Androgen receptor antagonist

SUMMARY:
RATIONALE: Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Androgens can cause the growth of prostate cancer cells. Drugs, such as goserelin, leuprolide, flutamide, or bicalutamide, may stop the adrenal glands from making androgens. Giving bortezomib with hormone therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving bortezomib with or without hormone therapy works in treating patients with relapsed prostate cancer.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate
* Relapsed disease after definitive local therapy, as documented only by a rise in prostate-specific antigen (PSA)

  * Experienced PSA relapse after definitive local therapy
  * Rising PSA (≥ 1.0 ng/mL after nadir < 1.0 ng/mL)

    * PSA increase of ≥ 0.3 ng/mL (increase occurred between 2 separate measurements taken ≥ 4 weeks apart)
  * The first of these two PSA values must rise above a previously recorded post-therapy nadir value
* Ineligible for curative therapy
* No clinical evidence of local recurrence (i.e., palpable induration or mass in the prostatic fossa) other than PSA elevation
* No evidence of palpable disease in the prostatic bed
* No metastatic disease (M0)

  * No non-nodal (> N1) metastasis
  * No evidence of osseous metastasis on bone scan within the past 28 days

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* ECOG 0-1

Life expectancy

* At least 1 year

Hematopoietic

* Platelet count ≥ 30,000/mm^3
* Absolute neutrophil count ≥ 1,000/mm^3

Hepatic

* No known hepatitis B or C positivity

Renal

* Creatinine clearance ≥ 30 mL/min

Immunologic

* No known human T-cell lymphotropic virus positivity
* No hypersensitivity to bortezomib, boron, or mannitol
* No known HIV 1 or 2 positivity
* No active, ongoing bacterial, viral, or fungal infection

Other

* Fertile patients must use effective contraception
* No peripheral neuropathy ≥ grade 2
* No other disease, condition, or social or geographic constraint that would preclude study participation
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* At least 6 months since prior hormonal therapy combined with radiation therapy as definitive therapy
* Neoadjuvant hormonal therapy prior to definitive therapy (e.g., surgery, radiation therapy, brachytherapy, or cryoablation) allowed
* No other concurrent hormonal therapy

Radiotherapy

* See Disease Characteristics
* More than 12 months since prior radioactive seed therapy
* No concurrent radiotherapy

Surgery

* See Disease Characteristics
* More than 4 weeks since prior surgery
* No concurrent surgery

Other

* No concurrent second-line herbal preparations, including PC-SPES
* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-10; Primary Completion 2009-10 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S. Kraft, MD, Principal Investigator — Medical University of South Carolina; Gustavo Leone, Study Chair — Medical University of South Carolina, Hollings Cancer Center
Locations (4):
- United States (4):
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A Only: Velcade: Patients who were enrolled to Part A but did not move on to Part B
- Part B (Velcade+LH-RH Antagonist+Adrogen Receptor): Patients who were enrolled only to part B.
- Part A + Part B: Patients who completed part A and moved in to Part B.
Period: Overall Study
Arm/Group | Part A Only: Velcade | Part B (Velcade+LH-RH Antagonist+Adrogen Receptor) | Part A + Part B
Started | 8 | 7 | 8
Completed | 8 | 7 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part B (Velcade + LH-RH Antagonist+Androgen Receptro: Patients who were enrolled only to part B
- Total: Total of all reporting groups
Arm/Group | Part A Only: Velcade | Part B (Velcade + LH-RH Antagonist+Androgen Receptro | Part A + Part B | Total
Number analyzed (Participants) | 8 | 7 | 8 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4 | 8
  >=65 years | 7 | 4 | 4 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 7 | 8 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 7 | 6 | 7 | 20
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Prostate-specific Antigen (PSA) Response
Time Frame: 3 months after the start of treatment
Measure: Number; unit: participants
Groups:
- Part A: Velcade: Patients who were enrolled to Part A but did not move on to Part B
- Part B: (Velcade+LH-RH Antagonist+Adrogen Receptor): Patients who were enrolled only to part B.
Arm/Group | Part A: Velcade | Part B: (Velcade+LH-RH Antagonist+Adrogen Receptor) | Part A + Part B
Number analyzed (Participants) | 8 | 7 | 8
participants | 1 | 6 | 5

2. Primary Outcome: Time to PSA Progression
Description: PSA progression is defined as a PSA increase of 50% over the nadir CR or CR/PR value on three successive PSA measurements two months apart to a value of >= 1.0 ng/ml.
Time Frame: From on study until time of PSA progression for up to two years
Population: Only patients with a CR were included in the analysis. No patients in Part A had a complete response. Time to progression for Part B only and Part A+Part B was calculated together. The information for the confidence interval is not available.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Part B and Part A + Part B: Patients who were enrolled to Part B (Velcade + LH-RH Antagonist+Androgen Receptor) and Part A (Velcade only) + Part B
Arm/Group | Part A Only: Velcade | Part B and Part A + Part B
Number analyzed (Participants) | 0 | 11
months |  | 5.49 [3.91 to NA] — NA is included to represent the value "infinity"

3. Secondary Outcome: Number of Patients Who Experienced an Adverse Event by CTCAE v. 2.0
Time Frame: From start of treatment until end of study, up to 6 months
Measure: Number; unit: participants
Groups:
- Part B (Velcade+Lh-RH Antagonist+ Androgen Receptor): patients who were enrolled only to Part B.
Arm/Group | Part A Only: Velcade | Part B (Velcade+Lh-RH Antagonist+ Androgen Receptor) | Part A + Part B
Number analyzed (Participants) | 8 | 7 | 8
participants | 8 | 7 | 8

4. Secondary Outcome: Disease-free Interval
Description: This will only be analyzed if sample size warrants the analysis.
Time Frame: 3 months after combined treatment
Population: data was not collected for this outcome measure.
Groups:
- Velcade and Hormonal Therapy: Patient will complete Part A (Velcade only). If the patient has a complete response, he will come off study. If the patient has progressive disease, he will start Velcade + Antiandrogen therapy. If the patient has a partial response or stable disease, he will start Velcade+antiandrogen after at least a 7-day break.
  After 3 months on Part B, if the patient has a complete response, he will come off study. Patients with a partial response or stable disease will repeat part B. Patients with progressive disease will come off study.
  Velcade: Part A: 1.3 mg/m2 administered on days 1, 4, 8 and 11 followed by 10 days rest. A second cycle will be given at the same schedule. Cycle 3 will include 3 weekly injections.
  Part B: 1.3mg/m2 administered weekly for 3 weeks followed by 1 week break
  LH-RH Agonist: given as a 3 month depo-injection
  Androgen Receptor Antagonists: given orally daily for 3 months
Arm/Group | Velcade and Hormonal Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: from start of treatment until end of study visit, about 6 months
Groups:
- Part A: Velcade Only: Patients who were enrolled to Part A but did not move on to Part B
Arm/Group | Part A: Velcade Only | Part B (Velcade+LH-RH Antagonist+Adrogen Receptor) | Part A + Part B
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 7/7 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: Velcade Only (N=8) | Part B (Velcade+LH-RH Antagonist+Adrogen Receptor) (N=7) | Part A + Part B (N=8)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Velcade Only (N=8) | Part B (Velcade+LH-RH Antagonist+Adrogen Receptor) (N=7) | Part A + Part B (N=8)
neuropathy (Nervous system disorders) | 8 | 0 | 8
fatigue (General disorders) | 8 | 5 | 6
anemia (Blood and lymphatic system disorders) | 5 | 0 | 7
thrombocytopenia (Blood and lymphatic system disorders) | 7 | 0 | 8
neutropenia (Blood and lymphatic system disorders) | 6 | 0 | 5
constipation (Gastrointestinal disorders) | 6 | 4 | 8
ileus (Gastrointestinal disorders) | 2 | 0 | 0
anorexia (General disorders) | 2 | 0 | 4
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
infection (Infections and infestations) | 1 | 0 | 1
vomiting (Gastrointestinal disorders) | 2 | 3 | 2
shingles (Infections and infestations) | 1 | 0 | 1
pain (General disorders) | 8 | 4 | 8
hypotension (Vascular disorders) | 1 | 1 | 2
dizziness (General disorders) | 3 | 1 | 1
insomnia (Psychiatric disorders) | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes